CLINICAL TRIAL: NCT03721315
Title: A Randomized Controlled Trial of Health Literacy Activation Among the Chronic Obstructive Pulmonary Disease Patients and Designated Support Dyad
Brief Title: Health Literacy Activation RCT Among the COPD Patients and Designated Support Dyad
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: SARS-CoV2 pandemic
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Audrey Djibo, Scientist, Interim Chair of the Research Division, Department of Medicine, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-19
Record Dates: First submitted 2018-10-23; First posted 2018-10-26 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: COPD Exacerbation
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group will receive the standard of care for this condition.
- Intervention (Experimental): This group will receive additional education along with their designated health support person prior to hospital discharge. This intervention does not include drugs/or devices.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — The health literacy enhancement will comprise of the following:
  * Practical day to day information to help manage the disease
  * Benefits of medication and adherence
  * Tips to improve managing shortness of breath
  * Proper use of inhalers (if applicable)
  * Managing daily activities
  Arms: Intervention

SUMMARY:
This study investigates whether increasing health literacy among COPD patients and their designated health coach during a hospital admission caused by symptoms exacerbation will lead to better health outcomes including increased health quality, and lower healthcare utilization.

DETAILED DESCRIPTION:
Until recently, contemporary methods to chronic disease management have failed to consistently tailor approaches among patients with low health literacy. They have produced mixed results in terms of successful interventions to address the needs of these populations. Low health literacy is especially common in medically underserved communities, including in North Philadelphia. This is reflected in the predominantly low-income and racial/ethnic minority population of the patients at this medical center. Management of chronic conditions such as COPD is complex. Patients with low health literacy find it especially challenging to self-navigate disease management. However, there is a lack of information on approaches to improve health outcomes among COPD patients with low health literacy.

The long-term goal is to develop and evaluate a model of interventions to improve healthcare outcomes for socially disadvantaged populations. The objective is to pilot a randomized controlled trial that evaluates the effects of an intervention that provides enhanced education and material support, on adherence to care, among patients admitted for COPD-related issues and their home support dyad.

The central hypothesis is that: compared to the standard educational intervention delivered by a registered nurse, the addition of an enhanced intervention (enhanced education, problem-solving skills and facilitative support) and the inclusion of a patient-designated support pair will result in greater adherence care and improves quality of life, especially among patients with low health literacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be 55 years old and above
* A history of hospital admissions for COPD related issues
* Able to designate a support person that can help them manage their condition
* Discharged home

Exclusion Criteria:

* Dyads unable to participate in the education session
* Patients discharged to a skilled nursing facility or rehabilitation facility.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-04-26 (Actual); Study Completion 2020-04-26 (Actual)

PRIMARY OUTCOMES:
Change in Respiratory Specific Health Related Quality of life (HRQoL) | 3 months
  Change in Respiratory Specific Health Related Quality of life (HRQoL) based on questionnaire responses at baseline and 3 months follow-up

SECONDARY OUTCOMES:
Medication adherence | 3 months
  Medication adherence measured by the number of prescription refills
Healthcare utilization | 3 months
  Healthcare utilization measured by the number of ER visits, and 30 day readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Djibo, PhD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Cross AJ, Thomas D, Liang J, Abramson MJ, George J, Zairina E. Educational interventions for health professionals managing chronic obstructive pulmonary disease in primary care. Cochrane Database Syst Rev. 2022 May 6;5(5):CD012652. doi: 10.1002/14651858.CD012652.pub2. PMID 35514131